CLINICAL TRIAL: NCT02187835
Title: Decreased EEG Complexity in Chronic Residual Schizophrenia
Brief Title: Decreased EEG Complexity in Schizophrenia
Status: Completed | Type: Observational
Sponsor: Uskudar University (Other)
Responsible Party: Principal Investigator, Gokben Hizli Sayar, M.D., Uskudar University
Other Study IDs: GHS001
Record Dates: First submitted 2014-07-09; First posted 2014-07-11 (Estimated); Last update posted 2014-07-11 (Estimated); Status verified 2014-07

CONDITIONS: Electrophysiological Randomness; Entropy
Keywords: complexity; electroencephalogram; entropy; negative symptoms; schizophrenia.
MeSH Terms: conditions — Schizophrenia

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (2):
- schizophrenia: patients with a diagnosis of schizohrenia
- control: healthy control group

SUMMARY:
Aim was to detect EEG complexity in a specific group of patients to contribute to the discussion whether schizophrenia is associated with increased or decreased complexity. We included the EEG recordings of patients with a diagnosis of schizophrenia. We hypothesized that chronic residual schizophrenia is characterized by decreased complexity in EEG.

DETAILED DESCRIPTION:
Twenty right-handed patients diagnosed with schizophrenia, residual subtype, by two senior psychiatrists according to the Diagnostic Statistical Manual of Mental Disorders 4th Edition (DSM-IV)were recruited from Neuropsychiatry Istanbul Hospital. Only patients scoring 4 or higher on the Clinical Global Impression Scale for Severity (CGI-S) were included. They were assessed with the Turkish version of the Positive and Negative Syndrome Scale. Data was collected with a 16-channel Neuroscan Synamps II (Neuroscan Products, Compumedics, Charlotte, NC, USA), silver-silver chloride electrodes were applied to the scalp surface according to the international 10-20 system

ELIGIBILITY:
Inclusion Criteria:

diagnosed with schizophrenia, residual subtype, by two senior psychiatrists according to the Diagnostic Statistical Manual of Mental Disorders 4th Edition (DSM-IV) were recruited from Neuropsychiatry Istanbul Hospital Only patients scoring 4 or higher on the Clinical Global Impression Scale for Severity (CGI-S)

Exclusion Criteria:

-

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: diagnosed with schizophrenia,
Sampling Method: Non-Probability Sample
Enrollment: 40 (Actual)
Dates: Start 2013-01; Primary Completion 2014-01 (Actual); Study Completion 2014-01 (Actual)

PRIMARY OUTCOMES:
the mean of the average Logarithmic Energy Entropy values | one day

SECONDARY OUTCOMES:
Hurst Exponent value | one day

CONTACTS AND LOCATIONS:
Locations (1):
- Uskudar University, NPIstanbul hospital, Istanbul, Umraniye, Turkey (Türkiye)

REFERENCES:
- See also: Neuropsychiatry Istanbul Hospital, Istanbul, Turkey — http://www.npistanbul.com